CLINICAL TRIAL: NCT04956289
Title: A Phase 2 Open-label Study to Assess the Safety, Tolerability, and Efficacy of Viltolarsen in Ambulant and Non-Ambulant Boys With Duchenne Muscular Dystrophy (DMD) Compared to Natural History Controls
Brief Title: Study to Assess the Safety, Tolerability, and Efficacy of Viltolarsen in Ambulant and Non-Ambulant Boys With DMD (Galactic53)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NS Pharma, Inc. (Industry)
Collaborators: Nippon Shinyaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS-065/NCNP-01-211
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-06

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — viltolarsen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Viltolarsen (Experimental): Patients amenable to exon 53 skipping will receive viltolarsen intravenous (IV) infusions, weekly, at 80 mg/kg for up to 48 weeks.
  Interventions: Drug: Viltolarsen

INTERVENTIONS:
Drug: Viltolarsen — Received during weekly intravenous infusions
  Other Names: NS-065/NCNP-01

SUMMARY:
This is a phase II, open-label study where weekly doses of 80 mg/kg viltolarsen is administered intravenously over a 48-week treatment period to ambulant and non-ambulant DMD patients over the age of 8 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (if age 18 years or older) or patient's parent(s) or legal guardian(s) has (have) provided written informed consent and Health Insurance Portability and Accountability Act authorization, where applicable, prior to any study-related procedures; patients younger than age 18 years will be asked to give written or verbal assent according to local requirements;
2. Patient has a confirmed diagnosis of DMD defined as:

   1. Patient is male with clinical signs compatible with DMD; and
   2. Patient has a confirmed DMD mutation(s) in the dystrophin gene that is amenable to skipping of exon 53 to restore the dystrophin messenger ribonucleic acid reading frame including determination of unambiguously defined exon boundaries (using techniques such as multiplex ligation-dependent probe amplification, comparative genomic hybridization array, or other techniques with similar capability);
3. Patient is more than 8 years of age at time of first infusion in the study;
4. Patient has a Brooke scale rating of 3 or better OR an upright FVC 30% or greater at Screening;
5. Patient, if sexually active, is willing to abstain from sexual intercourse or employ a barrier or medical method of contraception during and for 3 months following completion of IP administration;
6. Patient and patient's parent(s)/guardian(s) (if patient is <18 years of age) and/or caregiver(s) are willing and able to comply with scheduled visits, IP administration plan, and study procedures;
7. Patient must be on a stable dose of glucocorticoid (GC) or not treated with GC for at least 3 months prior to the first dose of IP and is expected to remain on stable dose of GC treatment or off GC for the duration of the study.

Other inclusion criteria may apply

Exclusion Criteria:

1. Patient has had an acute illness within 4 weeks prior to the first dose of IP;
2. Patient has evidence of symptomatic cardiomyopathy (New York Heart Association Class III or higher);
3. Patient requires ventilation support while awake during the day;
4. Patient has an allergy or hypersensitivity to IP or any of its constituents;
5. Patient has severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the investigator;
6. Patient has a previous or ongoing medical condition, medical history, physical findings, or laboratory abnormalities that could affect patient safety, make it unlikely that treatment and follow-up will be correctly completed, or impair the assessment of study results, in the opinion of the investigator;
7. Patient has had surgery within 3 months prior to the first anticipated administration of IP or has known plans to have surgery during the Treatment Period;
8. Patient has positive test results for hepatitis B antigen, hepatitis C antibody, or human immunodeficiency virus antibody at Screening;
9. Patient has been diagnosed with asthma that requires chronic treatment with a long-acting beta agonist;
10. Patient has relevant history of or current drug or alcohol abuse or use of any tobacco/marijuana products by smoking or vaping within 3 months prior to treatment with IP;
11. Patient is currently taking any other investigational drug or has taken any other investigational drug within 3 months prior to the first dose of IP or within 5 times the half-life of a medication, whichever is longer;
12. Patient has taken any gene therapy;
13. Patient is currently taking any other exon skipping agent or has taken any other exon skipping agent within 3 months prior to the first dose of IP;
14. Patient has hydronephrosis, hydroureter, renal or urinary tract calculi, or ureteral stenosis by renal ultrasound;
15. Patient was previously enrolled in an interventional study of viltolarsen.

Other exclusion criteria may apply

Min Age: 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-07-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Children's Hospital of Richmond at VCU, Richmond, Virginia, United States
- China (2):
  - The Third Medical Center of PLA General Hospital, Beijing
  - Hunan Children's Hospital, Changsha
- Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Roma, Italy
- Russia (2):
  - Russian National Research Medical University, Moscow
  - Saint Petersburg State Paediatric Medical University, Saint Petersburg
- Hospital Sant Joan de Deu, Barcelona, Spain
- Yeditepe University Kosuyolu Hospital, Istanbul, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study from July 1, 2021 to July 22, 2022 at 8 sites in the United States, Italy, Russia, Spain, and China.
Pre-assignment Details: A total of 27 participants were screened, but 3 participants did not meet inclusion or exclusion criteria and 4 participants failed to screen for other reasons.
Groups:
- Viltolarsen 80mg/kg: Participants who confirmed DMD with genetic deletions amenable to exon 53 skipping were administered an intravenous infusion of Viltolarsen 80 mg/kg once a week for up to 48 weeks.
Period: Overall Study
Arm/Group | Viltolarsen 80mg/kg
Started | 20
Ambulant | 10
Non-ambulant | 10
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The modified Intent-to-Treat (mITT) Population consisted of all patients who received at least 1 dose of IP and had a baseline assessment and at least 1 post-baseline efficacy assessment. This was the analysis population for the evaluation of efficacy. The Safety Population consisted of all patients who received at least 1 dose of IP. This was the primary analysis population for the evaluation of safety.
Arm/Group | Viltolarsen 80mg/kg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (5.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: No statistical analysis was performed for this endpoint. The information has been introduced in the section "Adverse Events".
Time Frame: baseline to up to 48 weeks of treatment
Population: The Safety Population consisted of all patients who received at least 1 dose of IP (Investigational Product). This was the primary analysis population for the evaluation of safety. It includes all patients treated with viltolarsen both ambulant (10) and non-ambulant (10).
Measure: Count of Participants; unit: Participants
Arm/Group | Viltolarsen 80mg/kg
Number analyzed (Participants) | 20
Participants | 19

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events by Maximum Severity
Description: as for outcome 1
Time Frame: baseline to up to 48 weeks of treatment
Population: The Safety Population consisted of all patients who received at least 1 dose of IP (Investigational Product). This was the primary analysis population for the evaluation of safety. It includes all patients treated with viltolarsen both ambulant (10) and non-ambulant (10). Only participants with Treatment-Emergent Adverse Events were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Viltolarsen 80mg/kg
Number analyzed (Participants) | 19
Participants
  Mild | 7
  Moderate | 12
  Severe | 0

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events by Highest Intervention Level Regarding Investigational Product
Description: as for outcome 1
Time Frame: baseline to up to 48 weeks of treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Viltolarsen 80mg/kg
Number analyzed (Participants) | 19
Participants
  Dose not changed | 16
  Dose reduced | 0
  Drug interrupted | 2
  Drug withdrawn | 0
  Not applicable | 1

4. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events by Worst Outcome
Description: as for outcome 1
Time Frame: baseline to up to 48 weeks of treatment
Population: The Safety Population consisted of all patients who received at least 1 dose of IP (Investigational Product). This was the primary analysis population for the evaluation of safety. It includes all patients treated with viltolarsen both ambulant (10) and non-ambulant (10). Only participants with Investigational Product-related Treatment Emergent Adverse Events were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Viltolarsen 80mg/kg
Number analyzed (Participants) | 19
Participants
  Recovered or resolved | 17
  Recovered or resolved with sequelae | 0
  Recovering or resolving | 0
  Not recovered or resolved | 2
  Fatal | 0

5. Primary Outcome: Number of Participants With Investigational Product-related Treatment Emergent Adverse Events
Description: as for outcome 1
Time Frame: baseline to up to 48 weeks of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Viltolarsen 80mg/kg
Number analyzed (Participants) | 20
Participants | 4

6. Primary Outcome: Number of Participants With Investigational Product-related Treatment Emergent Adverse Events by Maximum Severity
Description: as for outcome 1
Time Frame: baseline to up to 48 weeks of treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Viltolarsen 80mg/kg
Number analyzed (Participants) | 4
Participants
  Mild | 3
  Moderate | 1
  Severe | 0

7. Primary Outcome: Number of Participants With Investigational Product-related Treatment Emergent Adverse Events by Highest Intervention Level Regarding Investigational Product
Description: as for outcome 1
Time Frame: baseline to up to 48 weeks of treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Viltolarsen 80mg/kg
Number analyzed (Participants) | 4
Participants
  Dose not changed | 3
  Dose reduced | 0
  Drug interrupted | 1
  Drug withdrawn | 0

8. Primary Outcome: Number of Participants With Investigational Product-related Treatment Emergent Adverse Events by Worst Outcome
Description: as for outcome 1
Time Frame: baseline to up to 48 weeks of treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Viltolarsen 80mg/kg
Number analyzed (Participants) | 4
Participants
  Recovered or resolved | 4
  Recovered or resolved with sequelae | 0
  Recovering or resolving | 0
  Not recovered or resolved | 0
  Fatal | 0

9. Primary Outcome: Number of Participants With Adverse Event of Special Interest
Description: as for outcome 1
Time Frame: baseline to up to 48 weeks of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Viltolarsen 80mg/kg
Number analyzed (Participants) | 20
Participants | 5

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Description: Number of participants with Treatment Emergent Adverse Events as assessed by CTCAE v4.03
Arm/Group | Viltolarsen 80mg/kg
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 19/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viltolarsen 80mg/kg (N=20)
COVID-19 (Infections and infestations) | 6 (6)
Nasopharyngitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Influenza (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (13)
Food poisoning (Gastrointestinal disorders) | 2 (8)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Tension headache (Nervous system disorders) | 1 (2)
Pyrexia (General disorders) | 2 (3)
Gait inability (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Haematuria (Renal and urinary disorders) | 4 (6)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Protein urine (Investigations) | 1 (1)
Urine cytology abnormal (Investigations) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The most restrictive relevant agreement on the PI provides that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is not less than 30 days from the time submitted to the sponsor for review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT04956289/Prot_SAP_000.pdf